CLINICAL TRIAL: NCT01369225
Title: A Multicenter, Open-label Extension, Multiple Dose, Parallel Group Study To Investigate The Long-term Safety And Tolerability Of Aab-003 (Pf-05236812) Administered Intravenously In Subjects With Mild To Moderate Alzheimer's Disease Previously Treated With Aab-003 Or Placebo In Protocol B2601001
Brief Title: Open Label Extension Study Evaluating Safety and Tolerability of AAB-003 (PF-05236812) in Subject With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2601003
Record Dates: First submitted 2011-05-10; First posted 2011-06-08 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Randomized; Safety Study; Open Label
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.5 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 1 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 2 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 4 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 8 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)

INTERVENTIONS:
Drug: AAB-003 (PF-05236812) — 0.5 mg/kg AAB-003, IV
  Arms: 0.5 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 1 mg/kg AAB-003, IV
  Arms: 1 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 2 mg/kg AAB-003, IV
  Arms: 2 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 4 mg/kg AAB-003, IV
  Arms: 4 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 8 mg/kg AAB-003, IV
  Arms: 8 mg/kg AAB-003

SUMMARY:
This is a study to evaluate the safety and tolerability of multiple doses of AAB-003 (PF-05236812) in patients with mild to moderate Alzheimer's Disease. Patients who complete study B2601001 may participate in this trial and receive AAB-003 (PF-05236812). Each patient's participation will last approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of study B2601001
* MMSE 12 or greater

Exclusion Criteria:

* Study B2601001 Week 32 MRI with clinically important exclusionary findings.
* Experienced SAE, vasogenic edema and/or intracranial hemorrhage in study B2601001

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (15):
  - MD Clinical, Hallandale, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Trinity Care Solutions, Ocala, Florida
  - Advanced Imaging of Ocala, Ocala, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Foers Medical Arts Pharmacy, Bethesda, Maryland
  - CBH Health, LLC, Rockville, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - KNI Southwest Michigan Imaging Center, LLC, Kalamazoo, Michigan
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - DePaul Health Center-MRI Department, St Louis, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Central Jersey Radiology, Oakhurst, New Jersey
- South Korea (6):
  - Seoul National University Hospital, Department Neurology, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Department of Neurology, Incheon
  - Samsung Medical Center, Department of Neurology, Seoul
  - Korea University Anam Hospital IRB, Seoul
  - ASAN Medical Center, Seoul
  - Konkuk University Medical Center, Department of Neurology, Seoul

REFERENCES:
- [Derived] Delnomdedieu M, Duvvuri S, Li DJ, Atassi N, Lu M, Brashear HR, Liu E, Ness S, Kupiec JW. First-In-Human safety and long-term exposure data for AAB-003 (PF-05236812) and biomarkers after intravenous infusions of escalating doses in patients with mild to moderate Alzheimer's disease. Alzheimers Res Ther. 2016 Mar 1;8(1):12. doi: 10.1186/s13195-016-0177-y. PMID 26925577
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2601003&StudyName=Open%20Label%20Extension%20Study%20Evaluating%20Safety%20and%20Tolerability%20of%20AAB-003%20%28PF-05236812%29%20%20in%20Subject%20with%20Mild%20to%20Moderate%20Alzheimer%27s

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants who completed the first-in-human (FIH) study, B2601001.
Groups:
- AAB-003 0.5 mg/kg: Continued at same dose as preceding study B2601001 (NCT01369225), participants received intravenous (IV) infusion of AAB-003 (also known as PF-05236812) in a sterile vial at 0.5 mg/kg once every 13 weeks for up to 4 infusions.
- AAB-003 1 mg/kg: Continued at same dose as preceding study B2601001, participants received IV infusion of AAB-003 in a sterile vial at 1 mg/kg once every 13 weeks for up to 4 infusions.
- AAB-003 2 mg/kg: Continued at same dose as preceding study B2601001, participants received IV infusion of AAB-003 in a sterile vial at 2 mg/kg once every 13 weeks for up to 4 infusions.
- AAB-003 4 mg/kg: Continued at same dose as preceding study B2601001, participants received IV infusion of AAB-003 in a sterile vial at 4 mg/kg once every 13 weeks for up to 4 infusions.
- AAB-003 8 mg/kg: Continued at same dose as preceding study B2601001, participants received IV infusion of AAB-003 in a sterile vial at 8 mg/kg once every 13 weeks for up to 4 infusions.
- Placebo/AAB-003: Participants who received placebo in a preceding study B2601001 then received open-label active drug AAB-003. Subjects received either 0.5 mg/kg, 1 mg/kg, 2 mg/kg, 4mg/kg or 8 mg/kg once every 13 weeks for up to 4 infusions.
Period: Overall Study
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Started | 6 | 3 | 12 | 10 | 12 | 9
Completed | 4 | 3 | 9 | 8 | 10 | 9
Not Completed | 2 | 0 | 3 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Does Not Meet Entrance Criteria | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who were enrolled in the study and received at least 1 infusion of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003 | Total
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.5) | 63.0 (7.8) | 68.8 (10.6) | 71.3 (8.8) | 60.7 (5.8) | 71.7 (7.9) | 67.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 10 | 5 | 8 | 4 | 33
  Male | 2 | 1 | 2 | 5 | 4 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Week 52
Population: The safety analysis set included participants who received at least 1 infusion of study medication (including partial infusions).
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Number of Participants with AEs | 5 | 3 | 9 | 5 | 10 | 8
  Number of Participants with SAEs | 0 | 1 | 2 | 3 | 1 | 1

2. Primary Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, RBC morphology, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (coagulation panel, circulating immune complex, and complement activation).
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants | 3 | 2 | 8 | 7 | 10 | 6

3. Primary Outcome: Number of Participants With Potentially Clinically Important Vital Sign Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate <40 or >120 beats per minute (bpm); standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) of more than or equal to (>=)30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mmHg change from baseline in same posture or DBP <50 mm Hg.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Supine SBP <90 mm Hg | 1 | 0 | 0 | 0 | 0 | 1
  Supine DBP <50 mm Hg | 0 | 0 | 1 | 3 | 0 | 0
  Supine Pulse Rate <40 or >120 bpm | 0 | 0 | 0 | 0 | 1 | 0
  Supine SBP >=30 mm Hg Increase from Baseline | 3 | 1 | 1 | 2 | 4 | 1
  Supine DBP >=20 mm Hg Increase from Baseline | 2 | 1 | 4 | 5 | 1 | 2
  Supine SBP >=30 mm Hg Decrease from Baseline | 0 | 1 | 4 | 1 | 2 | 4
  Supine DBP >=20 mm Hg Decrease from Baseline | 0 | 1 | 5 | 3 | 3 | 5

4. Primary Outcome: Number of Participants With Potentially Clinically Important Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, QRS interval, and QT interval. Criteria for ECG changes meeting potential clinical concern included: PR interval >=300 milliseconds (msec) or >=25% increase when baseline is >200 msec and >=50% increase when baseline is less than or equal to (<=)200 msec; QRS interval >=200 msec or >=50% increase from baseline when baseline is less than or equal to 100 msec and >=25% increase when baseline is >100 msec; and QTcF >=450 msec or >=30 msec increase.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  PR Interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0
  QRS Complex >=200 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval 450 to <480 msec | 0 | 2 | 4 | 3 | 2 | 2
  QTcF Interval 480 to <500 msec | 0 | 0 | 1 | 1 | 1 | 0
  QTcF Interval >=500 msec | 0 | 0 | 1 | 0 | 0 | 0
  PR Interval >=25/50% Increase from Baseline | 0 | 0 | 0 | 0 | 0 | 0
  QRS Complex >=25/50% Increase from Baseline | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval >=30/<60 msec Change from Baseline | 2 | 1 | 4 | 4 | 1 | 2
  QTcF Interval >=60 msec Change from Baseline | 0 | 0 | 1 | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A full physical examination consisted of an examination of the abdomen, genitourinary and cardiovascular systems, lungs, lymph nodes, mouth, musculoskeletal and neurological systems, skin, extremities, head, ears, eyes, nose, throat and thyroid gland. Criteria for abnormal physical findings was based on the investigator's discretion and any new physical examination findings were documented as AEs. Only sites with at least 1 participant abnormality are reported.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Abdomen | 0 | 0 | 1 | 0 | 0 | 0
  Ears | 0 | 0 | 0 | 2 | 1 | 0
  Extremities | 0 | 0 | 0 | 0 | 0 | 1
  Eyes | 1 | 0 | 0 | 0 | 0 | 0
  General | 0 | 0 | 1 | 0 | 0 | 0
  Lymph Nodes | 0 | 1 | 0 | 0 | 0 | 0
  Musculoskeletal | 0 | 1 | 0 | 0 | 0 | 1
  Nose | 1 | 0 | 0 | 0 | 0 | 0
  Skin | 0 | 0 | 0 | 2 | 0 | 1
  Thyroid | 0 | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings
Description: Neurological examinations were done to the extent needed to assess the subject for any potential changes in neurological status, as determined by the investigator. Examinations included level of consciousness, speech, cranial nerves, motor, sensory, coordination, gait, and tendon reflexes. Only tests with at least 1 participant abnormality are reported.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Cranial Nerve Function | 1 | 0 | 0 | 2 | 0 | 0
  Coordination | 0 | 0 | 0 | 1 | 0 | 1
  Deep Tendon Reflexes | 0 | 0 | 1 | 0 | 0 | 0
  Motor Function | 0 | 1 | 0 | 0 | 0 | 1
  Gait and Station | 0 | 1 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. C-SSRS assesses whether participant experienced the following: completed suicide; suicide attempt; preparatory acts towards imminent suicidal behavior; suicidal ideation; self-injurious behavior, no suicidal intent. The results presented are the number of participants with completed suicide or non-fatal suicide events or behaviors. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0
  Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0
  Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0
  Suicidal Ideation | 0 | 0 | 1 | 0 | 1 | 0
  Self-Injurious Behavior, No Suicidal Attempt | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Any New Magnetic Resonance Imaging (MRI) Findings
Description: Brain MRIs were collected to assess for potential drug-related changes that might have constituted a safety concern. Findings suggestive of either vasogenic edema or intracranial hemorrhage were to be reported as AEs of special circumstance.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants | 1 | 1 | 0 | 0 | 0 | 1

9. Other Pre Specified Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer
Description: Number of participants with positive sample(s) in the ADA assay and in the neutralizing anti-drug antibodies (NAb) assay. An endpoint titer >=6.64 corresponded to positive ADA category value. The number of participants who tested positive on 1 or more occasions is reported.
Time Frame: Baseline, Week 52
Population: The safety analysis set included participants who received at least 1 infusion of study medication (including partial infusions); n=number of evaluable participants at the specified time point.
Measure: Number; unit: participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
participants
  Baseline (n=6,3,12,10,8) | 0 | 0 | 0 | 0 | 0 | 0
  Week 52 (n=4,3,9,8,10,8) | 0 | 0 | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Scores at Week 52
Description: ADAS-Cog is a structured scale that evaluates memory, orientation, attention, reasoning, language and constructional praxis. The ADAS-Cog comprises 11 items that are summed to a total score ranging from 0 to 70, with higher scores indicate greater cognitive impairment.
Time Frame: Baseline, Week 52
Population: The full analysis set included participants who were randomized and received at least 1 infusion of study medication; n=number of evaluable participants at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
units on a scale
  Baseline (n=6,3,12,10,12,9) | 12.0 (4.58) | 22.7 (11.79) | 25.1 (14.11) | 23.8 (9.21) | 19.6 (10.72) | 23.3 (11.00)
  Change at Week 52 (n=4,3,9,8,10,8) | 3.7 (3.98) | 3.0 (7.22) | 5.5 (4.30) | 2.8 (4.56) | 5.9 (4.22) | 2.5 (6.07)

11. Other Pre Specified Outcome: Change From Baseline in Disability Assessment in Dementia (DAD) at Week 52
Description: The DAD is a functional assessment comprised of 40 items (17 items related to self-care and 23 items involving instrumental activities of daily living). The DAD assessment is scored from 0 to 100; higher scores indicate better function.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
units on a scale
  Baseline (n=6,3,12,10,12,9) | 83.7 (12.50) | 73.3 (7.64) | 69.5 (23.82) | 72.4 (27.11) | 78.3 (19.48) | 81.1 (16.25)
  Change at Week 52 (n=4,3,9,8,10,9) | -5.0 (24.75) | -9.7 (6.43) | -10.4 (15.26) | -7.5 (6.72) | -5.2 (12.89) | -14.3 (20.51)

12. Other Pre Specified Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Behavioral Symptoms at Week 52
Description: The NPI is an instrument used to assess changes of behavior that have appeared in a defined period of time in subjects with Alzheimer's Disease and other dementias. Twelve behavioral areas are assessed: delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, nighttime behaviors, euphoria, appetite, and eating changes. The NPI score is based on frequency and severity of specific behaviors within these categories. Severity (1=Mild to 3=Severe), frequency (1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score (range 0-12). Total score=sum of each domain score (range 0-144); higher score=greater behavioral disturbances; negative change score from baseline=improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
units on a scale
  Baseline (n=6,3,12,10,12,9) | 11.2 (7.65) | 12.0 (13.45) | 7.1 (6.99) | 11.0 (16.73) | 9.6 (10.24) | 3.9 (3.92)
  Change at Week 52 (n=4,3,9,8,10,9) | -3.5 (4.36) | 5.7 (1.15) | 5.1 (8.39) | 4.5 (8.90) | 0.1 (12.54) | 13.9 (23.00)

13. Other Pre Specified Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) Scores at Week 52
Description: The CDR scale is a dementia staging instrument that tracks the progression of cognitive impairment in the following 6 categories: memory, orientation, judgment and problem solving, involvement in community affairs, home and hobbies, and personal care. The CDR-SB scale is obtained by summing the ratings in each of the 6 categories, ranging from 0 to 18. Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
units on a scale
  Baseline (n=6,3,12,10,12,9) | 9.00 (3.347) | 11.00 (1.000) | 11.33 (5.710) | 10.30 (4.473) | 10.33 (4.313) | 9.56 (3.941)
  Change at Week 52 (n=4,3,9,8,10,9) | 0.00 (0.816) | 0.33 (0.577) | 2.67 (2.291) | 2.38 (1.598) | 1.10 (2.378) | 2.56 (2.789)

14. Other Pre Specified Outcome: Change From Baseline in Mini-Mental State Exam (MMSE) Scores at Week 52
Description: The MMSE is a brief 30-point questionnaire test that is used to assess cognition. Scores range from 0 to 30, with higher scores indicating better cognitive state.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Number analyzed (Participants) | 6 | 3 | 12 | 10 | 12 | 9
units on a scale
  Baseline (n=6,3,12,10,12,9) | 24.7 (1.86) | 21.0 (4.36) | 19.3 (5.05) | 18.5 (4.86) | 21.3 (5.40) | 18.9 (5.64)
  Change at Week 52 (n=4,3,9,8,10,9) | -1.0 (2.94) | 1.7 (1.15) | -2.7 (2.78) | -2.1 (1.64) | -2.0 (2.16) | -1.7 (3.91)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and a non-serious event during the study.
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo/AAB-003
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/3 | 2/12 | 3/10 | 1/12 | 1/9
Other Adverse Events (participants affected / at risk) | 5/6 | 3/3 | 9/12 | 4/10 | 10/12 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AAB-003 0.5 mg/kg (N=6) | AAB-003 1 mg/kg (N=3) | AAB-003 2 mg/kg (N=12) | AAB-003 4 mg/kg (N=10) | AAB-003 8 mg/kg (N=12) | Placebo/AAB-003 (N=9)
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Device breakage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AAB-003 0.5 mg/kg (N=6) | AAB-003 1 mg/kg (N=3) | AAB-003 2 mg/kg (N=12) | AAB-003 4 mg/kg (N=10) | AAB-003 8 mg/kg (N=12) | Placebo/AAB-003 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal bruit (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Carotid bruit (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Parkinsonian gait (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Postural tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 3 | 2
Hypersexuality (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypnopompic hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Quadranopia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.